CLINICAL TRIAL: NCT01687712
Title: Phase III Investigator and Assessor Blinded 1:1 Randomized, Parallel-group Multicenter Study to Compare Efficacy and Safety of Two r-hFSH Formulations (AFOLIA vs Gonal-f® RFF) in Normal Ovulatory Women 35 to 42 Years Old Undergoing in Vitro Fertilization
Brief Title: Phase III Study Comparing Efficacy and Safety of AFOLIA vs Gonal-f® RFF in Women (35 to 42) Undergoing IVF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fertility Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIN3002
Record Dates: First submitted 2012-09-03; First posted 2012-09-19 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Infertility
Keywords: IVF; In vitro fertilization; Controlled ovarian stimulation; Follitropin; AFOLIA; Finox
MeSH Terms: conditions — Infertility | interventions — Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AFOLIA (Experimental): One subcutaneous injection of 225IU AFOLIA (follitropin alfa) per day (initial dose) for the first 5 days. From day 6 dose could be adjusted up (to a max of 450IU per day) or down (to a min of 75IU per day) in multiple increments of 37.5IU.
  Interventions: Drug: AFOLIA
- Gonal-f® RFF (Active Comparator): One subcutaneous injection of 225IU Gonal-f® RFF (follitropin alfa) per day (initial dose) for the first 5 days. From day 6 dose could be adjusted up (to a max of 450IU per day) or down (to a min of 75IU per day) in multiple increments of 37.5IU.
  Interventions: Drug: Gonal-f® RFF

INTERVENTIONS:
Drug: AFOLIA — 225IU subcutaneously, starting at the day of successful down-regulation for the first 5 days, followed by a treatment period with an increased dose until the point of ovulation induction has been reached
  Other Names: Follitropin-alfa
  Arms: AFOLIA
Drug: Gonal-f® RFF — 225IU subcutaneously, starting at the day of successful down-regulation for the first 5 days, followed by a treatment period with an increased dose until the point of ovulation induction has been reached
  Other Names: Follitropin-alfa
  Arms: Gonal-f® RFF

SUMMARY:
The purpose of this study is to show that AFOLIA, a recombinant manufactured human follicle stimulating hormone (r-hFSH) has a similar efficacy and safety profile compared to Gonal-f® RFF.

DETAILED DESCRIPTION:
Comparison of the clinical pregnancy rate in the AFOLIA group compared to the US approved Gonal-f® RFF Redi-ject group as the primary endpoint. Comparison of the number and size of follicles, the number of cycle cancellation, the hormone parameters and adverse events in the AFOLIA group compared to the Gonal-f® RFF group as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* 35 to 42 years of age
* Indication for controlled ovarian stimulation and IVF or intracytoplasmic sperm injection (ICSI)
* Regular menstrual cycles (25-35 days)
* History of a maximum of two fresh cycle treatments in the present series of assisted reproductive technologies (ART) at the day of first screening (thawed cycles are not subject to that criteria)
* Body mass index (BMI) ≥18 and ≤38 kg/m2
* Basal FSH <12 IU/L (cycle day 2-5)
* Antral follicle count (AFC) ≥ 10 to ≤20 follicles with a diameter of <11mm (sum of both ovaries) as measured on ultrasound (US) in the early follicular phase (menstrual cycle day 2-5)
* Documented history of infertility due to any of the following factors: tubal factor, mild endometriosis (American Society for Reproductive Medicine [ASRM] stage 1-2), male factor, unexplained infertility
* Presence of both ovaries by ultrasonography and normal uterine cavity (confirmed by hysterosalpingography, saline infusion sonography or hysteroscopy within 6 months before randomization)
* Male partner with semen analysis that is at least adequate for ICSI within 6 months prior to patient beginning down-regulation (invasive or surgical sperm retrieval, donor and/or cryopreserved sperm may be used)
* Willingness to participate in the study and to comply with the study protocol
* Signed informed consent prior to screening

Exclusion Criteria:

* Presence of pregnancy
* History of or active polycystic ovary syndrome (PCOS)
* AFC >20 follicles with a diameter of <11 mm (both ovaries combined) as measured on US in the early follicular phase (menstrual cycle day 2-5)
* History of >2 unsuccessful fresh ART retrieval cycles
* Presence of uncontrolled endocrine disorder
* Previous history or presence of severe OHSS
* Intrauterine fibroids ≥5 cm or otherwise clinically relevant pathology that could impair embryo implantation or pregnancy continuation
* History of recurrent spontaneous abortion (3 or more, even when unexplained)
* Presence of severe endometriosis (ASRM stage 3 or stage 4) or hydrosalpinx
* Neoplasia, including tumors of the hypothalamus and pituitary gland
* Abnormal bleeding of undetermined origin
* History of extrauterine pregnancy in the previous 3 months
* Known allergy or hypersensitivity to progesterone or to any of the excipients (including peanut oil) of the additional study medications (GnRH agonist, Ovidrel®, and Crinone 8%®)
* History of poor response to gonadotropin treatment (defined as fewer than 5 oocytes retrieved in a previous attempt)
* Any hormonal treatment within 1 month before the start of the FSH treatment, with the exception of levothyroxine)
* Egg donor
* Administration of other investigational products within the previous month
* Clinically abnormal findings at Visit 1
* Concomitant participation in another study protocol

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1100 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2015-09-10 (Actual); Study Completion 2016-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Jenkins, DM FRCOG, Study Director — Fertility Biotech AG
Locations (22):
- United States (22):
  - Physicians Research Group, Tempe, Arizona
  - HRC Fertility, Encino, California
  - Reproductive Associates of Delaware, Newark, Delaware
  - FL Fertility Institution, Tampa, Florida
  - Georgia Reproductive Specialists, Atlanta, Georgia
  - Fertility Centers of Illinois, Chicago, Illinois
  - In Via Fertility Specialists, Hoffman Estate, Illinois
  - Shady Grove Fertility RSC, Rockville, Maryland
  - Nevada Center for Reproductive Medicine, Reno, Nevada
  - Cooper Institute of Reproductive Hormonal Disorders, P.C., Marlton, New Jersey
  - Institute for Reproductive Health, Cincinnati, Ohio
  - Abington Reproductive Medicine, Abington, Pennsylvania
  - Main Line Fertility Center, Bryn Mawr, Pennsylvania
  - Shady Grove Fertility RSC, Chesterbrook, PA, Chesterbrook, Pennsylvania
  - University of Penn, Philadelphia, Pennsylvania
  - Fertility Associates of Memphis, Memphis, Tennessee
  - Texas Fertility Center, Austin, Texas
  - Center for Assisted Reproduction, Bedford, Texas
  - Fertility Specialists of Houston, Houston, Texas
  - Houston Fertility Institute, Houston, Texas
  - Center of Reproducitve Medicine, Webster, Texas
  - Jones Institute for Reproductive Medicine, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1548 subjects were enrolled, 1101 subjects were randomized and 1100 received Investigational Medicinal Product (IMP) at 22 investigational sites in the United States.
Pre-assignment Details: After the informed consent was signed, each subject received a subject identification number and underwent the down-regulation procedure. After a successful downregulation, subjects were centrally randomized in a 1:1 ratio to one of the treatment groups, AFOLIA or Gonal-f®RFF.
Period: Cycle 1
Arm/Group | AFOLIA | Gonal-f® RFF
Started | 549 | 551
Received hCG | 516 | 520
Oocyte/Ovum Pick Up | 513 | 517
Fertilization Performed | 508 | 512
Embryo Transfer | 466 | 483
Biochemical Pregnancy | 163 | 203
Clinical Pregnancy (Ascertained via an ultrasound scan.) | 114 | 138
Completed (A subject is listed as Completed if they delivered at least one live neonate.) | 101 | 122
Not Completed | 448 | 429
Not completed — Not Biochemically Pregnant | 386 | 348
Not completed — Early Pregnancy Loss | 43 | 60
Not completed — Ectopic Pregnancy | 5 | 5
Not completed — Heterotropic Pregnancy | 1 | 0
Not completed — Miscarriage/Spontaneous Abortion | 9 | 14
Not completed — Abortion | 3 | 0
Not completed — Intrauterine Fetal Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Cycle 2
Arm/Group | AFOLIA | Gonal-f® RFF
Started | 109 | 120
Received hCG | 107 | 119
Oocyte/Ovum Pick Up | 107 | 119
Fertilization Performed | 106 | 119
Embryo Transfer | 101 | 117
Biochemical Pregnancy | 35 | 43
Clinical Pregnancy (Ascertained via an ultrasound scan.) | 17 | 26
Completed (A subject is listed as Completed if they delivered at least one live neonate.) | 16 | 25
Not Completed | 93 | 95
Not completed — Not Biochemically Pregnant | 74 | 77
Not completed — Early Pregnancy Loss | 18 | 16
Not completed — Ectopic Pregnancy | 0 | 1
Not completed — Still Birth | 1 | 0
Not completed — Miscarriage/Spontaneous Abortion | 0 | 1
Period: Cycle 3
Arm/Group | AFOLIA | Gonal-f® RFF
Started | 28 | 24
Received hCG | 27 | 24
Ooctye/Ovum Pick-Up | 27 | 24
Fertilization Performed | 27 | 24
Embryo Transfer | 26 | 24
Biochemically Pregnant | 7 | 2
Clinical Pregnancy (Ascertained via an ultrasound scan.) | 5 | 0
Completed (A subject is listed as Completed if they delivered at least one live neonate.) | 4 | 0
Not Completed | 24 | 24
Not completed — Not Biochemically Pregnant | 21 | 22
Not completed — Early Pregnancy Loss | 1 | 2
Not completed — Ectopic Pregnancy | 1 | 0
Not completed — Miscarriage/Spontaneous Abortion | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intention to treat population, defined as all randomized subjects who received at least one dose of the study treatment, based on their randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | AFOLIA | Gonal-f® RFF | Total
Number analyzed (Participants) | 549 | 551 | 1100
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (2.16) | 37.8 (2.18) | 37.8 (2.17)
Age, Customized [Count of Participants; unit: Participants]
  35-37 | 275 | 276 | 551
  38-40 | 201 | 194 | 395
  41-42 | 73 | 81 | 154
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 549 | 551 | 1100
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 96 | 78 | 174
  Not Hispanic or Latino | 452 | 473 | 925
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 40 | 48 | 88
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 61 | 57 | 118
  White | 435 | 440 | 875
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 4 | 12
Height (m) [Mean (Standard Deviation); unit: meters] — Population: Number of subjects analysed is less than the number of subjects in the ITT population due to missing data.
  meters
    number analyzed (Participants) | 549 | 550 | 1099
    (all) | 1.643 (0.0660) | 1.642 (0.0684) | 1.642 (0.0672)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] — Population: Number of subjects analysed is less than the number of subjects in the ITT population due to missing data.
  kilograms
    number analyzed (Participants) | 541 | 546 | 1087
    (all) | 70.01 (13.803) | 71.12 (13.844) | 70.57 (13.828)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Population: Number of subjects analysed is less than the number of subjects in the ITT population due to missing data.
  kg/m^2
    number analyzed (Participants) | 541 | 545 | 1086
    (all) | 25.92 (4.738) | 26.38 (4.784) | 26.15 (4.765)
BMI Category (kg/m^2) [Count of Participants; unit: Participants]
  >=18 to <25 | 279 | 245 | 524
  >=25 to <30 | 150 | 184 | 334
  >=30 to <=38 | 109 | 112 | 221
  >38 | 3 | 4 | 7
  Unknown or Not Reported | 8 | 6 | 14
Primary Cause of Infertility [Count of Participants; unit: Participants] — Subjects can have more than one factor that causes infertility, therefore percentages may add up to more than 100.
  Participants
    Unexplained Infertility | 225 | 206 | 431
    Male Factor | 189 | 178 | 367
    Tubal Factor | 138 | 169 | 307
    Mild Endometriosis | 59 | 45 | 104
    Other | 28 | 41 | 69
Infertility Duration [Mean (Standard Deviation); unit: years] — Population: Number of subjects analysed is less than the number of subjects in the ITT population due to missing data.
  years
    number analyzed (Participants) | 548 | 550 | 1098
    (all) | 4.1 (4.61) | 4.2 (4.54) | 4.1 (4.58)
Number of previous fresh ART cycles [N(%)] [Count of Participants; unit: Participants] — Number of previous Assisted Reproductive Technology (ART) cycles a subject had prior to starting Cycle 1.
  Participants
    0 | 441 | 440 | 881
    1 | 81 | 77 | 158
    2 | 20 | 30 | 50
    ≥3 | 7 | 4 | 11
FSH at screening [Mean (Standard Deviation); unit: international units (IU)] — Measure of Follicle Stimulating Hormone (FSH) at screening. Population: Number of subjects analysed is less than the number of subjects in the ITT population due to missing data.
  international units (IU)
    number analyzed (Participants) | 548 | 550 | 1098
    (all) | 7.98 (4.636) | 7.76 (2.433) | 7.87 (3.700)
LH at screening [Mean (Standard Deviation); unit: international units (IU)] — Measure of Luteinizing Hormone (LH) at screening. Population: Number of subjects analysed is less than the number of subjects in the ITT population due to missing data.
  international units (IU)
    number analyzed (Participants) | 377 | 385 | 762
    (all) | 5.77 (3.36) | 5.74 (2.44) | 5.76 (2.93)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Pregnancy Rate After One Cycle of Treatment - ITT Population
Description: Clinical pregnancy was defined as presence of at least one intrauterine gestational sac and fetal heart activity as demonstrated by vaginal ultrasound at six weeks (42 +/- 1 day) post ET (Visit 11). The clinical pregnancy rate is the proportion of subjects who achieve clinical pregnancy, relative to the number of patients in the ITT population of the respective treatment arm.
Time Frame: Six weeks post embryo transfer
Population: Intention to treat population, defined as all randomized subjects who received at least one dose of study treatment, based on their randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 549 | 551
Participants
  Yes | 114 | 138
  No | 435 | 413
Statistical Analysis 1: Comparison: AFOLIA vs Gonal-f® RFF; The null and alternative hypotheses are as follows: H0: p2- p1 > ∆ and H1: p2- p1 ≤ ∆, where p1 is the clinical pregnancy rate in the AFOLIA treatment group, p2 is the clinical pregnancy rate in the Gonal f® treatment group, and Δ is the non-inferiority margin of 8%; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper limit of the two-sided 95% CI of the difference in pregnancy rates (Gonal-f® RFF - AFOLIA) did not exceed 8% (i.e. a one-sided hypothesis test at the 2.5% level of significance). The difference in rates (& Wald CI) was estimated using a logistic regression model with binomial distribution and identity link, with treatment and site as factors; Risk Difference (RD) = 3.7, 95% CI 2-sided [-1.3 to 8.7] — Note that "risk" in this context is the risk of clinical pregnancy. The difference is in the direction Gonal-f® RFF - AFOLIA

2. Primary Outcome: Clinical Pregnancy Rate After One Cycle of Treatment - PP Population
Description: Clinical pregnancy was defined as presence of at least one intrauterine gestational sac and fetal heart activity as demonstrated by vaginal ultrasound at six weeks (42 +/- 1 day) post ET (Visit 11). The clinical pregnancy rate is the proportion of subjects who achieve clinical pregnancy, relative to the number of patients in the PP population of the respective treatment arm.
Time Frame: Six weeks post embryo transfer
Population: Per-protocol population, defined as a subset of the ITT population composed of all patients without any major protocol deviation (i.e. one which would affect the primary efficacy endpoint assessment).
Measure: Count of Participants; unit: Participants
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 486 | 494
Participants
  Yes | 108 | 125
  No | 378 | 369
Statistical Analysis 1: Comparison: AFOLIA vs Gonal-f® RFF; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 2.8, 95% CI 2-sided [-2.5 to 8.1] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Exposure to r-hFSH Injections: Days of r-hFSH Stimulation - Cycle 1
Description: The number of days of r-hFSH stimulation a subject received during Cycle 1.
Time Frame: Measured at discretionary visits between Days 9 and 15 after FSH starts
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 549 | 551
days | 10.8 (1.72) | 11.0 (1.67)

4. Secondary Outcome: Exposure to r-hFSH Injections: Total Dose of r-hFSH (IU) - Cycle 1
Description: The total dose of r-hFSH that subjects received during Cycle 1.
Time Frame: Measured at discretionary visits between Days 9 and 15 after FSH starts.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: international unit (IU)
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 549 | 551
international unit (IU) | 3209.2 (1008.05) | 3343.6 (1005.08)

5. Secondary Outcome: Exposure to r-hFSH Injections: Daily Dose of r-hFSH (IU) - Cycle 1
Description: The mean dose of r-hFSH that subjects received in a day during Cycle 1.
Time Frame: Measured at discretionary visits between Days 9 and 15 after FSH starts.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: international unit (IU)
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 549 | 551
international unit (IU) | 292.1 (57.90) | 297.5 (56.97)

6. Secondary Outcome: Number of Oocytes Retrieved - Cycle 1
Description: The number of oocytes retrieved per subject, following hCG administration in Cycle 1.
Time Frame: Visit 8, 34-36 hours after hCG administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Oocytes retrieved
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 513 | 517
Oocytes retrieved | 11.3 (6.76) | 11.2 (6.63)
Statistical Analysis 1: Comparison: AFOLIA vs Gonal-f® RFF; The null and alternative hypotheses are as follows: H0: p2- p1 = 0 and H1: p2- p1 ≠0, where p1 is the least squares adjusted mean number of oocytes retrieved in the AFOLIA treatment group and p2 is the least squares adjusted mean number of oocytes retrieved in the Gonal f® treatment group; Test type: Superiority — Comparisons were tested against a null of zero at the two-side 5% significance level; p = 0.612, ANCOVA — P-values are based upon Type III sums of squares; Treatment group and Site are included as factors

7. Secondary Outcome: Local and Systemic Adverse Events: Dermal Response to Injection - Cycle 1
Description: Number of subjects reporting at least one dermal response to r-hFSH injection and number of subjects reporting no dermal responses.
Time Frame: Measure recorded in the Patient Diary which is maintained through entire FSH treatment, from FSH Start through to Day 16 after start of FSH (16 days).
Population: Safety population, defined as all randomized subjects who received at least one dose of study treatment, based on their randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 549 | 551
Participants
  Subjects who reported at least one dermal response | 37 | 42
  Subjects who reported no dermal responses | 512 | 509

8. Secondary Outcome: Local and Systemic Adverse Events: Dermal Response to Injection by Severity - Cycle 1
Description: Dermal response to r-hFSH injection as assessed by the investigator and categorized according to severity of reaction
Time Frame: Measure recorded in the Patient Diary which is maintained through entire FSH treatment, from FSH through to Day 16 after start of FSH (16 days).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 549 | 551
Participants
  No evidence of irritation | 28 | 25
  Minimal erythema, barely perceptible | 2 | 7
  Definited Erythema, readily visible; minimal edema | 0 | 1
  Definite Edema | 1 | 0

9. Secondary Outcome: Overall Summary of Adverse Events (AEs) - Cycle 1
Description: Summary of AEs, including the number of subjects experiencing to following during Cycle 1:
  At least one AE At least one treatment related AE At least one serious AE At least one AE leading to discontinuation of study drug At least one AE due to pregnancy complication
Time Frame: Measured from the start of FSH treatment through to either the end FSH treatment + 30 days (up to 46 days) or to the last Telephone Follow-up / Live Birth Questionnaire on pregnancy outcome (if applicable) (up to 10 months).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 549 | 551
Participants
  At least one AE | 403 | 391
  At least one treatment related AE | 202 | 197
  At least one serious adverse event | 32 | 31
  At least one AE leading to discontinuation | 2 | 1
  At least one AE due to pregnancy complication | 29 | 30

10. Secondary Outcome: Adverse Events of Special Interest: Ovarian Hyperstimulation Syndrome (OHSS) - Cycle 1
Description: Summary of the number of subjects with mild, moderate and severe OHSS. The total number of subjects with OHSS is also included.
Time Frame: Measured either 3 days after ooctye pick up (Visit 9) or 18 +/- 1 days after oocyte pick up (Visit 10).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 549 | 551
Participants
  Total Number of Subjects with OHSS | 13 | 12
  Number of Subjects with Mild OHSS | 6 | 4
  Number of Subjects with Moderate OHSS | 5 | 6
  Number of Subjects with Severe OHSS | 2 | 2

11. Secondary Outcome: Adverse Events of Special Interest: Ovarian Hyperstimulation Syndrome (OHSS) - Cycle 2
Description: as for outcome 10
Time Frame: Measured either 3 days after ooctye pick up (Visit 9) or 18 +/- 1 days after oocyte pick up (Visit 10).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 109 | 120
Participants
  Total Number of Subjects with OHSS | 1 | 3
  Number of Subjects with Mild OHSS | 1 | 1
  Number of Subjects with Moderate OHSS | 0 | 2
  Number of Subjects with Severe OHSS | 0 | 0

12. Secondary Outcome: Adverse Events of Special Interest: Ovarian Hyperstimulation Syndrome (OHSS) - Cycle 3
Description: as for outcome 10
Time Frame: Measured either 3 days after ooctye pick up (Visit 9) or 18 +/- 1 days after oocyte pick up (Visit 10).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 28 | 24
Participants
  Total Number of Subjects with OHSS | 0 | 0
  Number of Subjects with Mild OHSS | 0 | 0
  Number of Subjects with Moderate OHSS | 0 | 0
  Number of Subjects with Severe OHSS | 0 | 0

13. Secondary Outcome: Number of Subjects With Detectable Specific Serum Binding to FSH by Surface Plasmon Resonance - Cycle 1
Description: Measurement of the number of subjects with detectable specific serum binding to FSH by surface Plasmon resonance during Cycle 1.
Time Frame: Immunogenicity samples were taken at baseline, Visit 5 (8 days after start of treatment), Visit 9 (5 days after the end of FSH treatment), Visit 10 (18 +/- 1 days after oocyte retrieval), and Visit 11 (42 +/- 1 days after embryo transfer).
Population: Safety population, defined as all randomized subjects who received at least one dose of study treatment, based on their randomization. Percentages are based on the number of subjects in the safety population with data at the respective visit.
Measure: Count of Participants; unit: Participants
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 549 | 551
Participants
  Baseline | 1 | 1
  Visit 5: number analyzed (Participants) | 543 | 541
  Visit 5 | 1 | 1
  Visit 9: number analyzed (Participants) | 463 | 478
  Visit 9 | 1 | 1
  Visit 10: number analyzed (Participants) | 449 | 471
  Visit 10 | 1 | 1
  Visit 11: number analyzed (Participants) | 134 | 165
  Visit 11 | 0 | 1

14. Secondary Outcome: Number of Subjects With Detectable Specific Serum Binding to FSH by Surface Plasmon Resonance - Cycle 2
Description: Measurement of the number of subjects with detectable specific serum binding to FSH by surface Plasmon resonance during Cycle 2.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 109 | 120
Participants
  Baseline: number analyzed (Participants) | 107 | 120
  Baseline | 0 | 0
  Visit 5: number analyzed (Participants) | 108 | 120
  Visit 5 | 0 | 0
  Visit 9: number analyzed (Participants) | 101 | 115
  Visit 9 | 0 | 0
  Visit 10: number analyzed (Participants) | 101 | 114
  Visit 10 | 0 | 0
  Visit 11: number analyzed (Participants) | 19 | 32
  Visit 11 | 0 | 0

15. Secondary Outcome: Number of Subjects With Detectable Specific Serum Binding to FSH by Surface Plasmon Resonance - Cycle 3
Description: Measurement of the number of subjects with detectable specific serum binding to FSH by surface Plasmon resonance during Cycle 3.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 28 | 24
Participants
  Baseline | 0 | 0
  Visit 5: number analyzed (Participants) | 28 | 23
  Visit 5 | 0 | 0
  Visit 9: number analyzed (Participants) | 26 | 24
  Visit 9 | 0 | 0
  Visit 10: number analyzed (Participants) | 25 | 24
  Visit 10 | 0 | 0
  Visit 11: number analyzed (Participants) | 5 | 0
  Visit 11 | 0 | 0

ADVERSE EVENTS:
Groups:
- AFOLIA - Cycle 1: Enrolled subjects in Cycle 1 were randomized to one subcutaneous injection of 225IU AFOLIA (follitropin alfa) per day (initial dose) for the first 5 days. From day 6 dose could be adjusted up (to a max of 450IU per day) or down (to a min of 75IU per day) in multiple increments of 37.5IU.
- Gonal-f® RFF - Cycle 1: Enrolled subjects in Cycle 1 were randomized to one subcutaneous injection of 225IU Gonal-f (follitropin alfa) per day (initial dose) for the first 5 days. From day 6 dose could be adjusted up (to a max of 450IU per day) or down (to a min of 75IU per day) in multiple increments of 37.5IU.
- AFOLIA - Cycle 2: Enrolled subjects in Cycle 2 were randomized to one subcutaneous injection of 225IU AFOLIA (follitropin alfa) per day (initial dose) for the first 5 days. From day 6 dose could be adjusted up (to a max of 450IU per day) or down (to a min of 75IU per day) in multiple increments of 37.5IU.
- Gonal-f® RFF - Cycle 2: Enrolled subjects in Cycle 2 were randomized to one subcutaneous injection of 225IU Gonal-f (follitropin alfa) per day (initial dose) for the first 5 days. From day 6 dose could be adjusted up (to a max of 450IU per day) or down (to a min of 75IU per day) in multiple increments of 37.5IU.
- AFOLIA - Cycle 3: Enrolled subjects in Cycle 3 were randomized to one subcutaneous injection of 225IU AFOLIA (follitropin alfa) per day (initial dose) for the first 5 days. From day 6 dose could be adjusted up (to a max of 450IU per day) or down (to a min of 75IU per day) in multiple increments of 37.5IU.
- Gonal-f® RFF - Cycle 3: Enrolled subjects in Cycle 3 were randomized to one subcutaneous injection of 225IU Gonal-f (follitropin alfa) per day (initial dose) for the first 5 days. From day 6 dose could be adjusted up (to a max of 450IU per day) or down (to a min of 75IU per day) in multiple increments of 37.5IU.
Arm/Group | AFOLIA - Cycle 1 | Gonal-f® RFF - Cycle 1 | AFOLIA - Cycle 2 | Gonal-f® RFF - Cycle 2 | AFOLIA - Cycle 3 | Gonal-f® RFF - Cycle 3
All-Cause Mortality (participants affected / at risk) | 0/549 | 1/551 | 0/109 | 0/120 | 0/28 | 0/24
Serious Adverse Events (participants affected / at risk) | 32/549 | 31/551 | 2/109 | 6/120 | 3/28 | 0/24
Other Adverse Events (participants affected / at risk) | 403/549 | 391/551 | 69/109 | 66/120 | 13/28 | 12/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AFOLIA - Cycle 1 (N=549) | Gonal-f® RFF - Cycle 1 (N=551) | AFOLIA - Cycle 2 (N=109) | Gonal-f® RFF - Cycle 2 (N=120) | AFOLIA - Cycle 3 (N=28) | Gonal-f® RFF - Cycle 3 (N=24)
Foetal heart rate deceleration (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0
Accessory auricle (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cleft palate (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Congenital skin dimples (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cytogenetic abnormality (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Foetal chromosome abnormality (Congenital, familial and genetic disorders) | 1 | 3 | 0 | 0 | 0 | 0
Hypospadias (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mosaicism (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Polydactyly (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Trisomy 13 (Congenital, familial and genetic disorders) | 2 | 0 | 0 | 0 | 0 | 0
Trisomy 15 (Congenital, familial and genetic disorders) | 1 | 2 | 0 | 0 | 0 | 0
Trisomy 17 (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Trisomy 21 (Congenital, familial and genetic disorders) | 2 | 0 | 0 | 2 | 0 | 0
Trisomy 22 (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Trisomy 9 (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Turner's syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Death neonatal (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute fatty liver of pregnancy (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 5 | 0 | 0 | 0 | 0
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 1 | 0 | 0 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 1 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Heterotopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0 | 0 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 1 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 3 | 2 | 1 | 1 | 1 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 4 | 2 | 0 | 0 | 0 | 0
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Transverse presentation (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Vanishing twin syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 0 | 2 | 0 | 1 | 0 | 0 — Note: This includes subjects who were at risk of OHSS as well those who had actual OHSS.
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AFOLIA - Cycle 1 (N=549) | Gonal-f® RFF - Cycle 1 (N=551) | AFOLIA - Cycle 2 (N=109) | Gonal-f® RFF - Cycle 2 (N=120) | AFOLIA - Cycle 3 (N=28) | Gonal-f® RFF - Cycle 3 (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 1 | 0 | 0 | 0 | 0
Asthenopia (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 5 | 10 | 2 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 49 | 42 | 7 | 4 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 46 | 54 | 7 | 6 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 7 | 5 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 4 | 3 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 16 | 15 | 4 | 3 | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 13 | 10 | 4 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 8 | 9 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 3 | 11 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 53 | 55 | 8 | 11 | 0 | 2
Vomiting (Gastrointestinal disorders) | 11 | 14 | 1 | 1 | 0 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 3 | 0 | 0 | 0 | 0
Crying (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 13 | 14 | 2 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 6 | 8 | 1 | 1 | 0 | 0
Injection site erythema (General disorders) | 82 | 76 | 11 | 5 | 2 | 0
Injection site haematoma (General disorders) | 3 | 2 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Injection site inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 2 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 7 | 7 | 1 | 0 | 0 | 0
Injection site scab (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 8 | 4 | 0 | 0 | 0 | 0
Injection site vesicles (General disorders) | 3 | 4 | 0 | 0 | 0 | 0
Irritability (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 2 | 2 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 4 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 1 | 1 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 3 | 2 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infected bites (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 9 | 6 | 1 | 1 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Salpingitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 4 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 3 | 1 | 1 | 0 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 39 | 36 | 8 | 12 | 3 | 3
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 | 3 | 0 | 0 | 0 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 15 | 15 | 2 | 2 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 105 | 89 | 13 | 11 | 3 | 2
Procedural vomiting (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 0 | 0 | 0
Blood oestrogen increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Infertility tests (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 21 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 16 | 0 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 0 | 0
Aphonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 10 | 7 | 2 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 3 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 145 | 127 | 14 | 16 | 2 | 5
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 7 | 1 | 1 | 1 | 0
Migraine with aura (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Retinal migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 4 | 2 | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abortion early (Pregnancy, puerperium and perinatal conditions) | 43 | 60 | 18 | 16 | 1 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 7 | 9 | 0 | 1 | 1 | 0
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 4 | 0 | 1 | 1 | 0
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 4 | 0 | 0 | 0 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Subchorionic haematoma (Pregnancy, puerperium and perinatal conditions) | 2 | 5 | 0 | 0 | 0 | 0
Subchorionic haemorrhage (Pregnancy, puerperium and perinatal conditions) | 3 | 1 | 0 | 0 | 0 | 0
Vanishing twin syndrome (Pregnancy, puerperium and perinatal conditions) | 1 | 6 | 0 | 0 | 0 | 0
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 3 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 1 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Emotional disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 7 | 4 | 1 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 4 | 3 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 2 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Adnexa uteri pain (Reproductive system and breast disorders) | 7 | 3 | 1 | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 0 | 1 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 12 | 8 | 0 | 2 | 0 | 0
Cervical discharge (Reproductive system and breast disorders) | 2 | 0 | 0 | 1 | 0 | 0
Cervical polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Coital bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 4 | 3 | 0 | 0 | 0 | 0
Fallopian tube cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypomenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 2 | 0 | 0 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ovarian enlargement (Reproductive system and breast disorders) | 3 | 1 | 0 | 0 | 0 | 0
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 16 | 12 | 3 | 2 | 0 | 0 — Note: This includes subjects who were at risk of OHSS as well those who had actual OHSS.
Pelvic discomfort (Reproductive system and breast disorders) | 8 | 10 | 1 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 6 | 0 | 0 | 0 | 0
Uterine cervix stenosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0
Uterine pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 1 | 1 | 0 | 0 | 0
Uterine spasm (Reproductive system and breast disorders) | 8 | 9 | 2 | 2 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 2 | 4 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 14 | 19 | 1 | 2 | 1 | 0
Vaginal odour (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 4 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 2 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 15 | 2 | 0 | 0 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 2 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 2 | 0 | 0 | 0 | 0 | 0
Sinus operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
Uterine dilation and curettage (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Diastolic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 11 | 8 | 1 | 3 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contract agreement. Results may not be published or referred to, in whole or in part, without the prior express written consent of the Sponsor.